CLINICAL TRIAL: NCT02885324
Title: Pilot Study of Cabozantinib for Recurrent or Progressive Central Nervous System Tumors in Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to meet accrual goals.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Scott Coven, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0601
Record Dates: First submitted 2016-08-24; First posted 2016-08-31 (Estimated); Results first posted 2022-08-15 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Malignant Brain Tumor; High Grade Glioma
Keywords: High Grade Glioma; Cabozantinib; GBM; Children; AA
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Brain Neoplasms; Glioma | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Cabozantininb will be taken daily at a dose of 40 mg/m2. Drug cycles will last 28 days and be continuous for up to 12 months of therapy on study.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Subjects will receive Cabozantinib
  Other Names: XL 184; Cabometyx

SUMMARY:
This pilot will study the feasibility and exploratory efficacy of using Cabozantinib for recurrent or refractory central nervous system tumors for which there are no curative options. Patients will also be followed for safety, time to progression, event free survival and overall survival

ELIGIBILITY:
Inclusion Criteria

1. Age: Patients must be ≥2 years and ≤21 years of age
2. Diagnosis: Patients with relapsed or refractory central nervous system tumors. Patients must have had histological verification of malignancy at original diagnosis or relapse. Metastatic disease to the spine or primary tumors in the spine are eligible. Patients may be in first, second, or third relapse. Subjects with intrinsic brain stem gliomas may be eligible with or without histological confirmation. Please contact study chair prior to enrollment.
3. Disease Status: Patients must have measurable disease. Linear enhancement of leptomeningeal without measurable mass is excluded.
4. Therapeutic Options: Patient's current disease state must be one for which there is no accepted standard therapy, no known curative therapy or therapy proven to prolong survival with an acceptable quality of life. For patients in whom surgery is feasible, maximal surgical resection must have occurred.
5. Performance Level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age (See Appendix 1). Note: Neurologic deficits in patients must have been relatively stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
6. Subjects must have a reasonable life expectancy of at least 2 months.
7. Prior Therapy

   a. Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy i. Cytotoxic chemotherapy (including investigational agents) or biologic agents (eg. Cytokines or antibodies): At least 3 weeks after the last dose.

   ii. Nitrosoureas/mitomycin C: At least 6 weeks from the last dose. iii. XRT: At least 14 days after local palliative XRT (small port); At least 150 days must have elapsed if prior TBI, craniospinal XRT or if ≥ 50% radiation of pelvis; At least 42 days must have elapsed if other substantial BM radiation. e.g. Stem cell Infusion without TBI: No evidence of active graft vs. host disease and at least 56 days must have elapsed after transplant or stem cell infusion.
8. Organ Function Requirements:

   a. Adequate bone marrow function defined as: absolute neutrophil count (ANC ≥1000/mm3) i. Platelet count ≥ 100,000/ mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) ii. Patients with bone marrow metastatic disease will not be eligible. b. Adequate renal function defined as: i. Creatinine clearance or radioisotope GFR ≥ 70mL/min/1.73 m² or a serum creatinine based on age/gender as follows:

   Age Maximum Serum Creatinine (mg/dL) Male Female 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

   ≥ 16 years 1.7 1.4 The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

   ii. Urine protein: ≤ 30 mg/dL in urinalysis or ≤ 1+ on dipstick, unless quantitative protein is < 1000 mg in a 24 hour urine sample.

   c. Adequate Liver Function Defined as:

   i. Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age ii. SGPT (ALT) ≤ 110 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.

   iii. Serum albumin ≥ 2.8 g/dL. d. Adequate coagulation status defined as: PT and INR ≤ 1.5x ULN e. Adequate pancreatic function defined as: Serum amylase and lipase ≤ 1.5 x ULN f. Adequate blood pressure control defined as: A blood pressure (BP) ≤ the 95th percentile for age, height and gender (Appendix II) despite optimal antihypertensive treatment within 7 days of the first dose of the study treatment. Please note that 3 serial blood pressures should be obtained and averaged to determine baseline BP.

   g. Central nervous system function defined as: Patients with seizure disorder may be enrolled if receiving non-enzyme inducing anticonvulsants and well controlled. See Appendix III for a list of recommended non-enzyme inducing anticonvulsants.

   h. Adequate cardiac function defined as: i. No history of congenital QTc syndrome, NYHA Class III or IV congestive heart failure (CHF) ii. No clinical significant cardiac arrhythmias, stroke or myocardial infarction within 6 months prior to enrollment iii. QTc

   ≤ 480 msec. Note: One ECG must be performed for eligibility determination. If the QTc is > 480 msec, two additional ECGs must be performed and the average of the three ECGs will be used to determine eligibility. Patients with Grade 1 prolonged QTc (450-480 msec) at the time of study enrollment should have correctable causes of prolonged QTc addressed if possible (i.e. electrolytes, medications). See Appendix IV for a list of drugs that prolong QTc.
9. Informed consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate will be obtained according to institutional guidelines.
10. Archival tumor tissue slides must be sent or available, except for patients with intrinsic pontine glioma meeting the remainder of the inclusion criteria.

Exclusion Criteria

1. Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogentic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two methods of birth control- a medically accepted barrier method of contraceptive method (e.g., male or female condom) and a second effective method of birth control- during protocol therapy and for at least 4 months after the last dose of cabozantinib. Abstinence is an acceptable method of birth control.
2. Concomitant Medications:

   1. Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible.
   2. Investigational drugs: Patients who are currently receiving another investigational drug are not eligible.
   3. Anti-cancer agents: patients who are currently receiving other anti-cancer agents are not eligible.
   4. CYP3A4 active agents: Patients must not be receiving any of the following potent CYP3A4 inducers or inhibitors: erythromycin, clarithromycin, ketoconazole, azithromycin, itraconazole, grapefruit juice or St. John's wort. A list of other known CYP3A4 inducers and inhibitors that should be discontinued prior to initiation of protocol therapy and should be avoided during study therapy if reasonable alternatives exist is included in Appendix V.
   5. Patients who are receiving systemic therapeutic treatment anticoagulation are not eligible. Patients receiving prophylactic systemic anticoagulation will be allowed with heparin or LMWH as long as eligibility PT/INR requirements are met. Concomitant anticoagulation with oral anticoagulations (e.g. warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg. Clopidogrel) are not allowed.
   6. Enzyme-inducing anticonvulsants: Patients must not have received enzyme-inducing anticonvulsants within 14 days prior to enrollment (See Appendix III for a list of unacceptable enzyme inducing anticonvulsants).
   7. QTc Agents: Patients who are receiving drugs that prolong QTc are not eligible (See Appendix IV for a list of agents).
3. Patients must be able to swallow intact tablets. Patients who cannot swallow intact tablets are not eligible.
4. Patients with active bleeding are not eligible. Specifically, no clinically significant GI bleeding, GI perforation, intra-abdominal abscess or fistula for 6 months prior to enrollment, no hemoptysis or other signs of pulmonary hemorrhage for 3 months prior to enrollment.
5. Patients with evidence of an acute intracranial or intratumoral hemorrhage on CT or MRI are not eligible (patients with evidence of resolving hemorrhage will be eligible).
6. Major surgery within 28 days of enrollment. Complete wound healing from major or minor surgery must have occurred prior to enrollment. Minor surgery (including uncomplicated tooth extractions) within 7 days of enrollment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible;
7. Concurrent uncontrolled hypertension defined as sustained blood pressure>95% for age, height and gender (systolic or diastolic) despite optimal antihypertensive treatment within 7 days of the first dose of study treatment.
8. Patients with any medical or surgical conditions that would interfere with gastrointestinal absorption of this oral agent are not eligible.
9. Infection: Patients who have an uncontrolled infection are not eligible.
10. Patients who have received a prior solid organ transplantation are not eligible.
11. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
12. Subjects who have received cabozantinib or have an allergy to cabozantinib are excluded. Subjects who have previously received tyrosine kinase inhibitors are allowed.
13. Subjects who have not received radiation therapy as part of their prior treatment are excluded.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Coven, DO, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Response
Description: To assess the number of participants with best response of CR, PR, SD or PD. Response criteria are assessed based on the product of the longest diameter and its longest perpendicular diameter.
  Complete response (CR): Disappearance of all target lesions Partial response (PR): ≥50% decrease in the sum of the products of the two perpendicular diameters of all target lesions (up to 5), taking as reference the initial baseline measurements Stable disease (SD): Neither sufficient decrease in the sum of the products of the two perpendicular diameters of all target lesions to qualify for PR, nor sufficient increase in a single target lesion to qualify for PD.
  Progressive Disease (PD): The appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Overall Survival
Description: To assess the number of participants who survived at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 4
Participants | 2

3. Secondary Outcome: Number of Participants With Progression Free Survival
Description: To assess the number of participants who had progression free survival at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=4)
Hypothyroidism (Endocrine disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Hepatobiliary disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Hepatobiliary disorders) | 2
Blood bilirubin increased (Hepatobiliary disorders) | 1
Blurred vision (Eye disorders) | 1
Confusion (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Depressed level of consciousness (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dry eye (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysarthria (Psychiatric disorders) | 1
Dysgeusia (General disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphasia (Psychiatric disorders) | 1
Epistaxis (Blood and lymphatic system disorders) | 1
diplopia (Eye disorders) | 1
right visual field deficit (Eye disorders) | 1
Fatigue (General disorders) | 3
Gait disturbance (General disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (General disorders) | 2
Hemoglobin increased (Blood and lymphatic system disorders) | 1
Hemorrhoids (General disorders) | 1
jaundice (Hepatobiliary disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypoxia (General disorders) | 1
stubbed toe (Injury, poisoning and procedural complications) | 1
Intracranial hemorrhage (General disorders) | 1
Laryngeal inflammation (Musculoskeletal and connective tissue disorders) | 1
Lipase increased (General disorders) | 1
Memory impairment (Psychiatric disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
unable to coordinate movements (Nervous system disorders) | 1
Pain in extremity (Injury, poisoning and procedural complications) | 2
Palmar-plantar erythrodysethesia syndrome (Skin and subcutaneous tissue disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
respiratory secretions (Respiratory, thoracic and mediastinal disorders) | 1
subject hospitalized in acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Serum amylase increased (General disorders) | 1
hair color change (Skin and subcutaneous tissue disorders) | 2
Skin infection (Skin and subcutaneous tissue disorders) | 1
Somnolence (General disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Voice alteration (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight loss (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT02885324/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT02885324/ICF_001.pdf